CLINICAL TRIAL: NCT02562170
Title: Protexa® Versus TiLoopBra® in Immediate Breast Reconstruction- A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daphne Gschwantler-Kaulich, Ass.Prof.Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1401/2013
Record Dates: First submitted 2015-09-18; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer; Hereditary Breast and Ovarian Cancer Syndrome
Keywords: breast; reconstruction; mesh; acellular dermal matrix
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TiLoop Bra (Active Comparator): immediate breast reconstruction with an implant and TiLoop Bra
  Interventions: Device: TiLoop Bra
- Protexa (Active Comparator): immediate breast reconstruction with an implant and Protexa
  Interventions: Device: Protexa

INTERVENTIONS:
Device: TiLoop Bra
  Arms: TiLoop Bra
Device: Protexa
  Arms: Protexa

SUMMARY:
Randomized controlled trial to look at early complications, cosmetic outcome, patient satisfaction and thickness of the tissue overlying the implant at the lower pole in immediate implant based breast reconstruction after Skin or Nipple Sparing Mastectomy with either a mesh (TiLOOP Bra) or an ADM (Protexa). Multicenter austrian trial with four breast cancer centers, 50 patients randomized 1:1 in the TiLoop or Protexa group.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients with indication for skin or nipple sparing mastectomy
* BRCA1/2 mutation carriers with indication for skin or nipple sparing mastectomy

Exclusion Criteria:

* prior local radiotherapy
* inflammatory breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
complications | up to two weeks after surgery
  hematoma, seroma, infection, skin necrosis, capsular contracture, implant loss
change of baseline patient quality of life after 3 and 6 months | up to two weeks after surgery (=baseline), 3 and 6 months after surgery
  questionnaire
change of baseline cosmetic outcome after 3 and 6 months | up to two weeks after surgery (=baseline), 3 and 6 months after surgery
  four point Harris Scale (1=poor, 4=excellent)
change of baseline thickness of the tissue overlying the implant at the lower pole after 3 and 6 months | up to two weeks after surgery (=baseline), 3 and 6 months after surgery
  The thickness of the tissue covering the implant in the lower pole im mm measured by ultrasound
complications | 3 months after surgery
  hematoma, seroma, infection, skin necrosis, capsular contracture, implant loss
complications | 6 months after surgery
  hematoma, seroma, infection, skin necrosis, capsular contracture, implant loss

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Gschwantler-Kaulich, Ass.Prof.Dr., Principal Investigator — Medical University Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Gschwantler-Kaulich D, Schrenk P, Bjelic-Radisic V, Unterrieder K, Leser C, Fink-Retter A, Salama M, Singer C. Mesh versus acellular dermal matrix in immediate implant-based breast reconstruction - A prospective randomized trial. Eur J Surg Oncol. 2016 May;42(5):665-71. doi: 10.1016/j.ejso.2016.02.007. Epub 2016 Feb 23. PMID 26947961